CLINICAL TRIAL: NCT07244042
Title: Effects of Modified Constraint-induced Movement Therapy With and Without Proprioceptive Neuromuscular Facilitation Techniques on Upper Extremity Function in Pediatric Stroke Patients
Brief Title: Effects of Modified CIMT With and Without PNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/MAIDA SHABBIR
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Stroke
Keywords: Modified CIMT; Proprioceptive Neuromuscular Facilitation(PNF); Pediatric Stroke
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized clinical trial over an intervention period of six-week. 20 pediatric stroke patients with upper extremity impairments will be randomly assigned to two groups: one receiving modified CIMT alone and the other receiving modified CIMT combined with PNF techniques. Pre- and post-intervention assessments will be conducted using standardized measures, such as Pediatric Motor Activity Log(PMAL) for upper extremity function, Modified Ashworth Scale(MAS) and Manual Ability Classification System(MACS). Muscle tone and physical activity status will also be evaluated. Data will be entered and analyzed in SPSS V-26.0 to compare improvements in motor function between the two groups, with statistical significance assessed to determine the efficacy of each intervention.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Intervention Group (Modified CIMT+PNF) (Active Comparator): Modified CIMT: Constraining the unaffected arm with a mitt or splint to encourage use of the affected arm (3-5 times a week).
  PNF Techniques: Includes rhythmic initiation, combination of isotonics, and replication exercises to enhance proprioception and motor control in the affected arm (10 reps of each technique for 15-20 minutes with rest interval) Rest Interval for 1-2 minute to prevent fatigue Routine Physiotherapy Exercises: Targeted exercises focusing on strength, range of motion, and coordination.
  * Strengthening: 3 sets of 10-12 reps per targeted muscle group (e.g., biceps, wrist extensors).
  * Range of Motion (ROM): 10-15 repetitions per joint (e.g., shoulder, elbow, wrist).
  * Coordination and Functional Training: Structured tasks such as reaching and grasping toys or objects for 15-20 minutes.
  Duration: 6 weeks
  Interventions: Other: Modified CIMT; Other: Proprioceptive Neuromuscular Facilitation
- Group B: Control Group (Modified CIMT only) (Active Comparator): Warm-Up Exercises:
  10-15 minutes of light exercises for the affected arm, focusing on gentle range of motion.
  Modified CIMT: Constraining the unaffected arm with a mitt or splint to promote use of the affected arm(3-5 times a week). Routine Physiotherapy Exercises: Targeted exercises focusing on strength, range of motion, and coordination.
  * Strengthening: 3 sets of 10-12 reps per targeted muscle group (e.g., biceps, wrist extensors).
  * Coordination and Functional Training: Structured tasks such as reaching and grasping toys or objects for 15-20 minutes.
  Duration: 6 week
  Interventions: Other: Modified CIMT

INTERVENTIONS:
Other: Modified CIMT — Modified CIMT Protocol: Participants wear a mitt on the unaffected hand daily for 5 hours approximately to encourage the use of the affected upper limb. They engage in task-oriented activities designed to improve motor function, hand-eye coordination, and strength of the affected extremity.
Other: Proprioceptive Neuromuscular Facilitation — PNF (Proprioceptive Neuromuscular Facilitation) is a stretching and rehabilitation technique that combines muscle contraction and relaxation with passive stretching to improve flexibility, range of motion, and muscle control
  Arms: Group A: Intervention Group (Modified CIMT+PNF)

SUMMARY:
This randomized clinical trial investigates the effects of modified CIMT with and without the addition of PNF techniques on upper extremity function in pediatric stroke patients, aiming to determine whether combining these approaches yields superior motor recovery.This study will be conducted as a randomized clinical trial over an intervention period of six-week. 20 pediatric stroke patients with upper extremity impairments will be randomly assigned to two groups: one receiving modified CIMT alone and the other receiving modified CIMT combined with PNF techniques. Pre- and post-intervention assessments will be conducted using standardized measures, such as Pediatric Motor Activity Log(PMAL) for upper extremity function, Modified Ashworth Scale(MAS) and Manual Ability Classification System(MACS). Muscle tone and physical activity status will also be evaluated. Data will be entered and analyzed in SPSS V-26.0 to compare improvements in motor function between the two groups, with statistical significance assessed to determine the efficacy of each intervention

DETAILED DESCRIPTION:
Pediatric stroke often results in impaired upper extremity function, significantly affecting children's ability to perform daily tasks and reducing their overall quality of life. Traditional therapeutic approaches may not provide sufficient recovery, necessitating the exploration of more effective interventions. Constraint-Induced Movement Therapy (CIMT) has been shown to improve motor function in pediatric stroke patients by enhancing the use of the affected limb. However, incorporating Proprioceptive Neuromuscular Facilitation (PNF) techniques may enhance the outcomes further by stimulating neuromuscular pathways to improve strength and coordination. The objective of this study is to compare the effects of modified CIMT with and without the addition of PNF techniques on upper extremity function in pediatric stroke patients, aiming to determine whether combining these approaches yields superior motor recovery.

This study will be conducted as a randomized clinical trial over an intervention period of six-week. 20 pediatric stroke patients with upper extremity impair-ents will be randomly assigned to two groups: one receiving modified CIMT alone and the other receiving modified CIMT combined with PNF techniques. Pre- and post-intervention assessments will be conducted using standardized measures, such as Pediatric Motor Activity Log(PMAL) for upper extremity function, Modified Ashworth Scale(MAS) and Manual Ability Classification System(MACS). Muscle tone and physical activity status will also be evaluated. Data will be entered and analyzed in SPSS V-26.0 to compare improvements in motor function between the two groups, with statistical significance assessed to determine the efficacy of each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Paeds Patients with confirmed diagnosis of Stroke
* Children between age 5 to 13 years
* Modified Ashworth Scale spasticity level 1 and 2.
* Patients having Manual Ability Classification System Score between 3 to 6.
* GMFCS level 1 and 2
* Patient having in affected upper extremity at least 20◦ of active wrist extension starting from the full flexion, 10◦ of active extension or abduction in the thumb, and 10◦ of active extension in the metacarpophalangeal and interphalangeal joints of the other fingers

Exclusion Criteria:

* Patients with epilepsy or seizure disorder
* Patients with history of botulinum toxin injection, cognitive impairment, fracture and any surgical procedure in upper extremity

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Pediatric Motor Activity Log (PMAL) | Base line, 3rd Week, 6th week
  This log will be used to assess the spontaneous use of the affected upper limb in daily activities. Parents/guardians will rate the frequency and quality of use.
Modified Ashworth Scale (MAS) | Base line, 3rd Week, 6th week
  This scale will be used to assess the degree of spasticity in the affected upper limb.
Manual Ability Classification System (MACS) | Base line, 3rd Week, 6th week
  The MACS will classify the participant's ability to handle objects and perform manual tasks in daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Maida Shabbir, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saygili F, Guclu-Gunduz A, Eldemir S, Eldemir K, Ozkul C, Gursoy GT. Effects of modified-constraint induced movement therapy based telerehabilitation on upper extremity motor functions in stroke patients. Brain Behav. 2024 Jun;14(6):e3569. doi: 10.1002/brb3.3569. PMID 38873866
- [Background] Adiguzel H, Kirmaci ZIK, Gogremis M, Kirmaci YS, Dilber C, Berktas DT. The effect of proprioceptive neuromuscular facilitation on functional skills, muscle strength, and trunk control in children with cerebral palsy: A randomized controlled trial. Early Hum Dev. 2024 May;192:106010. doi: 10.1016/j.earlhumdev.2024.106010. Epub 2024 Apr 15. PMID 38653163